CLINICAL TRIAL: NCT02568384
Title: Open Label, Single-center Study of the Onyx Meter and App System for Blood Glucose Monitoring in Insulin-Dependent and Insulin-using, Non-Insulin-Dependent Diabetes Mellitus Patients to Demonstrate Usability in a Clinical Setting.
Brief Title: Evaluation of an Ascensia Blood Glucose Meter and App System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCA-2014-006-01
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Results first posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Users of Onyx BG Meter / App System (Experimental): Subjects with diabetes used the Onyx Blood Glucose (BG) Meter / App System at home. The enrollment goal for the intended use population:
  1. 40 to 70% of subjects will have type 1 diabetes
  2. Not more than 30% of subjects will use an insulin pump
  Interventions: Device: Onyx BG Meter / App System

INTERVENTIONS:
Device: Onyx BG Meter / App System — Subjects with diabetes used the Onyx BG Meter / App System at home and assessed software operations, ease of use of the system, and clarity and utility of user instructions.

SUMMARY:
The purpose of this study is to assess the usability of the Onyx system in the hands of subjects with Insulin Dependent Diabetes Mellitus (IDDM) or insulin-using subjects with Non-IDDM.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18-75 years, male or female
* Read and understand English
* Have diagnosis of type 1 or insulin-using type 2 diabetes for at least 6 months
* Be taking multiple daily injections (MDI) of at least two pre-meal bolus injections daily or using an insulin pump
* Performing self-monitoring of blood glucose at home at least twice daily
* Have an iOS mobile device or Android mobile device with blue tooth capability
* iOS device: iPod or iPhone 5 or later version with iOS 8.0 software or higher (no tablets)
* Android: smart phone, 4.4 version and higher (no tablets)
* Be willing to utilize the ONYX App on personal mobile device which communicates to meter to manage diabetes (including use of the bolus calculator)
* Be ambulatory and have transportation to the study site

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Pregnancy
* Physical, visual or neurological impairments that would make the person unable to perform testing with the BGM
* Working for a competitive medical device company, or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company.
* A condition, which in the opinion of the investigator or designee, would put the person or study conduct at risk (reason for exclusion will be clearly documented by investigator or designee on the subject disposition form).
* Proliferative retinopathy or history of retinal laser surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute Inc.
Locations (1):
- AMCR Institute, Escondido, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Users of Onyx BG Meter / App System: Subjects with diabetes used the Onyx BG Meter / App System at home. The enrollment goal for the intended use population:
  1. 40 to 70% of subjects will have type 1 diabetes
  2. Not more than 30% of subjects will use an insulin pump
  Onyx BG Meter / App System: Subjects with diabetes used the Onyx BG Meter / App System at home and assessed software operations, ease of use of the system, and clarity and utility of user instructions.
Period: Overall Study
Arm/Group | Users of Onyx BG Meter / App System
Started | 45
Completed | 43
Not Completed | 2
Not completed — Mobile devices incompatible with App | 2

BASELINE CHARACTERISTICS:
Arm/Group | Users of Onyx BG Meter / App System
Number analyzed (Participants) | 45
Age, Continuous [Mean (Full Range); unit: years] | 45.9 [19 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Percent of Responses From Persons Who Performed Each "Software Operations" Task and Rated Each Statement as Strongly Agree, Agree, or Neither Agree Nor Disagree.
Description: For "software operations" tasks, subjects rated statements about software operations tasks as 1Strongly Agree, 2Agree, 3Neither Agree nor Disagree, 4Disagree, 5Strongly Disagree, or 6No opinion. Software operations tasks included:
  * Obtain a synced blood glucose reading
  * Initiation and use of insulin bolus calculator
  * Access and interpret glucose displays such as expanded graph (modal day) and sequential views.
Time Frame: 3 weeks
Population: While 43 subjects completed the questionnaire, responses with 'No opinion' were not counted in the total used to calculate percent of responses for each statement.
Measure: Number; unit: Percent of Responses
Groups:
- Users of Onyx BG Meter / App System: Subjects with diabetes used the Onyx BG Meter / App System at home.
  Onyx BG Meter / App System: Subjects with diabetes used the Onyx BG Meter / App System at home and assessed software operations, ease of use of the system, and clarity and utility of user instructions.
Arm/Group | Users of Onyx BG Meter / App System
Number analyzed (Participants) | 43
Percent of Responses
  I could successfully sync my BG reading with App | 95.4
  I could successfully initiate/use Bolus Calculator | 89.7
  I could access/interpret displays in the App. | 95.4

2. Secondary Outcome: Percent of Responses From Persons With Diabetes That Rated Ease of Use For Onyx Glucose Meter and App System as Either Very Simple or Simple or Neither Simple Nor Difficult
Description: Staff obtained responses from persons with diabetes using short questionnaires to provide feedback on the basic operation of the Onyx Glucose Meter and App System. Subjects could respond '1Very Simple' or '2Simple' or '3Neither Simple nor Difficult' or '4Difficult' or '5Very Difficult' or '6No Opinion'.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Responses
Arm/Group | Users of Onyx BG Meter / App System
Number analyzed (Participants) | 43
Percentage of Responses
  Accessing the Expanded Graph view was: | 97.6
  Accessing the My Readings view was: | 97.7
  Using the My Readings view was: | 100
  Using the Edit view was: | 97.6
  Using the Meal Marker Selection screen was: | 97.5
  I am satisfied w how easily meter BG syncs w App. | 90.7

3. Secondary Outcome: Percent of Responses From Persons With Diabetes That Either 'Strongly Agree' or 'Agree' or Are 'Neither Agree Nor Disagree' With Questionnaire Statements Regarding Clarity and Utility of User Instructions For Onyx Glucose Meter and App System
Description: Staff obtained responses from persons with diabetes using short questionnaires to provide feedback on the clarity and utility of user instructions for the Onyx Glucose Meter and App System. Subjects could respond '1Strongly Agree' or '2Agree' or '3Neither Agree nor Disagree' or '4Disagree' or '5Strongly Disagree' or '6No Opinion'.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of responses <or = 3
Arm/Group | Users of Onyx BG Meter / App System
Number analyzed (Participants) | 43
percentage of responses <or = 3
  The User Guide was helpful in using Onyx system.: number analyzed (Participants) | 34
  The User Guide was helpful in using Onyx system. | 100
  The Quick Reference Guide was helpful.: number analyzed (Participants) | 33
  The Quick Reference Guide was helpful. | 100
  The App Help section was helpful in using Onyx.: number analyzed (Participants) | 32
  The App Help section was helpful in using Onyx. | 100

4. Other Pre Specified Outcome: HbA1c% From Study Start to End of Study
Description: Laboratory reports were used to compare HbA1c results from subjects at visit 1 with HbA1c results at Visit 2 (end of study).
Time Frame: 3 weeks
Population: Change in %HbA1c.
Measure: Mean (Full Range); unit: %HbA1c
Arm/Group | Users of Onyx BG Meter / App System
Number analyzed (Participants) | 43
%HbA1c
  Study Visit 1 | 8.04 [5.7 to 11.9]
  Study Visit 2 | 7.78 [5.7 to 12.0]

5. Other Pre Specified Outcome: Average Change in Subject Fructosamine From Study Start to End of Study
Description: Laboratory reports were used to compare Fructosamine results from subjects at visit 1 with Fructosamine results at Visit 2 (end of study).
Time Frame: 3 weeks
Population: Change in umol/L
Measure: Mean (Full Range); unit: umol/L
Arm/Group | Users of Onyx BG Meter / App System
Number analyzed (Participants) | 43
umol/L
  Study Visit 1 | 331.5 [230 to 533]
  Study Visit 2 | 312.3 [206 to 525]

6. Other Pre Specified Outcome: Average Change in Subject Body Weight From Study Start to End of Study
Description: Subject Body Weight results at visit 1 were compared with Body Weight results at Visit 2 (end of study).
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: pounds
Arm/Group | Users of Onyx BG Meter / App System
Number analyzed (Participants) | 43
pounds
  Study Visit 1 | 189.5 [107 to 297]
  Study Visit 2 | 190.0 [108 to 294]

7. Other Pre Specified Outcome: Average Change in Total Daily Insulin Dose From Study Start to End of Study
Description: Subjects' self-reported Total Daily Insulin Doses at visit 1 were compared with their self-reported Total Daily Insulin Doses at Visit 2 (end of study).
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: insulin units
Arm/Group | Users of Onyx BG Meter / App System
Number analyzed (Participants) | 43
insulin units
  Study Visit 1 | 58.6 [10 to 162]
  Study Visit 2 | 61.5 [10 to 234]

ADVERSE EVENTS:
Arm/Group | Users of Onyx BG Meter / App System
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days